CLINICAL TRIAL: NCT01999257
Title: Assessing the Outcomes of Web-based Pre-test Educational Module for Carrier Genetic Screening in Individuals of Ashkenazi Jewish Descent
Brief Title: Efficacy Study of an Online Educational Module Before Carrier Genetic Screening in Persons of Ashkenazi Jewish Descent.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Guillaume Sillon, Genetic counsellor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 3281
Record Dates: First submitted 2013-11-25; First posted 2013-12-03 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Tay Sachs Disease; Canavan Disease; Familial Dysautonomia
Keywords: Genetic Counseling; Technology; Ashkenazi Jewish; Carrier screening
MeSH Terms: conditions — Tay-Sachs Disease; Canavan Disease; Dysautonomia, Familial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- In-person counselling (No Intervention): Similar to standard of care, wherein Ashkenazi Jewish individuals seeking carrier genetic screening meet a genetic counsellor for an in-person education and counselling session.
- Online pre-test genetic education tool (Active Comparator): Use of a web-based pre-test education program, wherein the information from a typical genetic counselling session for carrier screening in Ashkenazi Jewish individuals is presented.
  Interventions: Other: Online pre-test genetic education tool

INTERVENTIONS:
Other: Online pre-test genetic education tool — See Arm Descriptions above.
  Arms: Online pre-test genetic education tool

SUMMARY:
The investigators have developed a new website to educate persons of Ashkenazi Jewish ancestry about their increased risk for having children with certain genetic conditions, and the genetic testing the investigators offer. This study aims to pilot the website to find out whether it is effective and to learn what the investigators can improve.

Participants in the study will be assigned to one of two conditions:

1. Standard in-person genetic counselling session to learn about inheritance of Ashkenazi Jewish genetic conditions and genetic testing. Participants will fill out two short questionnaires, one before and one after the genetic counselling session. They will then be given a requisition form to undergo blood draw for genetic testing at the Montreal General Hospital test centre.
2. Use of a web-based pre-test genetic counselling tool to learn about inheritance of Ashkenazi Jewish genetic conditions and genetic testing. They will fill out two short questionnaires, one before, and one after using the web-based tool. They will then be electronically sent a requisition form to undergo blood draw for genetic testing at the Montreal General Hospital test centre.

In both conditions, genetic test results will be communicated by telephone once they are available. Participants' genetic test results will not be used in any way for the study.

DETAILED DESCRIPTION:
In Montreal, individuals of Ashkenazi Jewish descent are eligible to have carrier screening for three genetic conditions: Tay-Sachs disease, Canavan disease, and familial dysautonomia. The investigators have developed a new website to educate persons of Ashkenazi Jewish ancestry about their increased risk for having children with these genetic conditions, and the genetic testing the investigators offer. This study aims to pilot the website to find out whether it is effective and to learn what the investigators can improve. Specifically, the investigators will measure knowledge acquisition, level of anxiety, and degree of satisfaction with their experience.

Participants in the study will be assigned to one of two conditions:

1. Standard in-person genetic counselling session to learn about inheritance of Ashkenazi Jewish genetic conditions and genetic testing. Participants will fill out two short questionnaires, one before and one after the genetic counselling session. These questionnaires assess demographic information, knowledge regarding the three genetic conditions listed above, feelings and anxiety levels, e-health literacy, and overall satisfaction. They will then be given a requisition form to undergo blood draw for genetic testing at the Montreal General Hospital test centre.
2. Use of a web-based pre-test genetic counselling tool to learn about inheritance of Ashkenazi Jewish genetic conditions and genetic testing. They will fill out two short questionnaires, one before, and one after using the web-based tool. These questionnaires are similar to those in the condition above, except there will also be questions regarding the utility of the web-based tool and ways to improve the tool. Participants will then be electronically sent a requisition form to undergo blood draw for genetic testing at the Montreal General Hospital test centre.

In both conditions, genetic test results will be communicated by telephone once they are available. Participants' genetic test results will not be used in any way for the study.

ELIGIBILITY:
Inclusion Criteria:

* At least one grandparent of Ashkenazi Jewish descent
* Access to computer at home and computer literate

Exclusion Criteria:

* Participant or participant's partner is pregnant at time of study
* Family history of an Ashkenazi Jewish genetic condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-04 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Knowledge of Ashkenazi Jewish genetic conditions | 1 hour
  Evaluated by questionnaire developed specifically for this study.

SECONDARY OUTCOMES:
Patient anxiety | 1 hour
  Evaluated by 6-item short form state trait anxiety inventory (Becker and Marteau 1992)
Satisfaction with web-based/in-person genetic counselling | 1 hour
  Assessed by questionnaire, developed from pre-existing genetic counselling research (Shiloh et al. 1990; Yip et al. 2003)
Perceived risk of having a child with an Ashkenazi Jewish genetic condition | 1 hour
  Evaluated by questionnaire developed specifically for this study.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Sillon, MSc, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal General Hospital (MUHC), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Publication of study results in a peer-reviewed journal.